CLINICAL TRIAL: NCT01015287
Title: A Comparison of Prasugrel at the Time of Percutaneous Coronary Intervention (PCI) Or as Pretreatment At the Time of Diagnosis in Patients With Non-ST-Elevation Myocardial Infarction (NSTEMI): The ACCOAST Study
Brief Title: A Comparison of Prasugrel at PCI or Time of Diagnosis of Non-ST Elevation Myocardial Infarction
Acronym: ACCOAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12918; H7T-MC-TADF (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes; Heart Disease; Percutaneous Coronary Intervention; P2Y12; NSTEMI
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Diseases; Non-ST Elevated Myocardial Infarction | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non pre-treatment (Experimental): A placebo oral loading dose is given at the time of diagnosis and a 60 milligrams (mg) oral loading dose of prasugrel is given at the time of PCI followed by 5 mg or 10 mg oral daily maintenance dose of prasugrel for 30 days.
  Interventions: Drug: Placebo; Drug: Prasugrel
- Split Loading Dose (Experimental): A 30 mg oral loading dose of prasugrel is given at diagnosis and a 30 mg oral dose of prasugrel is given at the time of PCI followed by 5 mg or 10 mg oral daily maintenance dose of prasugrel for 30 days
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Placebo — Administered once orally
  Arms: Non pre-treatment
Drug: Prasugrel — Administered orally
  Other Names: LY640315; Efient; Effient; CS-747

SUMMARY:
The purpose of this trial is to investigate the potential benefits/risks regarding pretreatment with prasugrel in non-ST-elevation myocardial infarction (NSTEMI) participants with elevated troponin scheduled for coronary angiography/percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
This trial consists of two arms. One arm is a non pre-treatment arm. Participants in this arm will receive placebo immediately after NSTEMI diagnosis and prior to the diagnostic coronary angiography. A 60 mg prasugrel loading dose will be given immediately after coronary angiography when proceeding to PCI. Subsequently, participants will receive daily maintenance doses of prasugrel until day 30. Participants who are greater than or equal to 75 years of age or who have a body weight less than 60 kilograms (kg) will receive 5 mg oral dose daily. All others will receive a 10 mg oral daily maintenance dose for 30 days.

The other arm is a pre-treatment arm where participants will receive a split loading dose regimen with 30 mg of prasugrel administered immediately after NSTEMI diagnosis and prior to diagnostic coronary angiography. The remainder of the loading dose (30 mg) will be administered when the participants are proceeding to PCI. Subsequently, participants will receive daily maintenance doses of prasugrel until day 30. Participants who are greater than or equal to 75 years of age or who have a body weight less than 60 kg will receive 5 mg oral dose daily. All others will receive a 10 mg oral daily maintenance dose for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Have acute coronary syndrome consisting of non-ST-segment elevation with elevated troponin
* Scheduled for coronary angiography/PCI greater than or equal to 2 and less than 24 hours from time of planned randomization, but no more than 48 hours from randomization
* Must be eligible for treatment with prasugrel, aspirin (ASA), and a glycoprotein IIb/IIIa receptor (GPIIb/IIIa) inhibitor as per respective labels
* May be on a maintenance dose of clopidogrel 75 mg and must be able to switch to prasugrel
* Must be enrolled at a cardiac catheterization laboratory hospital or at a hospital/ambulance service affiliated with a cardiac catheterization laboratory hospital

Exclusion Criteria:

* Present with ST-segment elevation myocardial infarction (STEMI) at the time of entry or randomization
* Have cardiogenic shock
* Have refractory ventricular arrhythmias
* Have New York Heart Association (NYHA) Class IV congestive heart failure (CHF)
* Have had cardiac arrest within 1 week of entry or randomization into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4033 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (153):
- Austria (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Braunau am Inn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Belgium (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bonheiden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bruges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleroi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yvoir
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saskatoon, Saskatchewan
- Czechia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hradec Králové
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olomouc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pilsen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ústí nad Labem
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku, Finland
- France (25):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bastia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bron
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caluire-et-Cuire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cannes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Châteauroux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corbeil-Essonnes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lagny-sur-Marne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Le Coudray
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metz-Tessy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montauban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreuil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pierre-Bénite
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vannes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villeurbanne
- Germany (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Nauheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Segeberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bonn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dachau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eutin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kassel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludwigshafen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rastatt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostock
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villingen-Schwenningen
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Balatonfüred
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pécs
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zalaegerszeg
- Israel (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beer Yaakov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nahariya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tiberias
- Italy (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arezzo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chieti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grosseto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Legnano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lucca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Massa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pavia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perugia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prato
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reggio Emilia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Udine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Venezia
- Latvia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liepāja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riga
- Lithuania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klaipedos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilnius
- Netherlands (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eindhoven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeuwarden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nieuwegein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zwolle
- Poland (25):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bełchatów
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chrzanów
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grodzisk Mazowiecki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kłodzko
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mielec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nałęczów
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nowy Sącz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nowy Targ
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nysa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ostrowiec Świętokrzyski
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oświęcim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Polanica-Zdrój
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Puławy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Radom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sanok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stalowa Wola
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Starogard Gdański
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tarnów
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wejherowo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Portugal (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Braga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carnaxide
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Faro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leiria
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Slovakia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Banská Bystrica
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nitra
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg, Sweden
- Turkey (Türkiye) (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antalya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fatih
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Isparta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kayseri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kocaeli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Şişli

REFERENCES:
- [Derived] Silvain J, Rakowski T, Lattuca B, Liu Z, Bolognese L, Goldstein P, Hamm C, Tanguay JF, Ten Berg J, Widimsky P, Miller D, Portal JJ, Collet JP, Vicaut E, Montalescot G, Dudek D; ACCOAST Investigators. Interval From Initiation of Prasugrel to Coronary Angiography in Patients With Non-ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol. 2019 Mar 5;73(8):906-914. doi: 10.1016/j.jacc.2018.11.055. PMID 30819358
- [Derived] Porto I, Bolognese L, Dudek D, Goldstein P, Hamm C, Tanguay JF, Ten Berg J, Widimsky P, Le Gall N, Zagar AJ, LeNarz LA, Miller D, Montalescot G; ACCOAST Investigators. Impact of Access Site on Bleeding and Ischemic Events in Patients With Non-ST-Segment Elevation Myocardial Infarction Treated With Prasugrel: The ACCOAST Access Substudy. JACC Cardiovasc Interv. 2016 May 9;9(9):897-907. doi: 10.1016/j.jcin.2016.01.041. PMID 27151605
- [Derived] Dudek D, Dziewierz A, Widimsky P, Bolognese L, Goldstein P, Hamm C, Tanguay JF, LeNarz L, Miller DL, Brown E, Ten Berg J, Montalescot G; ACCOAST Investigators. Impact of prasugrel pretreatment and timing of coronary artery bypass grafting on clinical outcomes of patients with non-ST-segment elevation myocardial infarction: From the A Comparison of Prasugrel at PCI or Time of Diagnosis of Non-ST-Elevation Myocardial Infarction (ACCOAST) study. Am Heart J. 2015 Nov;170(5):1025-1032.e2. doi: 10.1016/j.ahj.2015.07.017. Epub 2015 Jul 26. PMID 26542513
- [Derived] Widimsky P, Motovska Z, Bolognese L, Dudek D, Hamm C, Tanguay JF, Ten Berg J, Brown E, LeNarz L, Miller DL, Montalescot G; ACCOAST Investigators. Predictors of bleeding in patients with acute coronary syndromes treated with prasugrel. Heart. 2015 Aug;101(15):1219-24. doi: 10.1136/heartjnl-2015-307686. Epub 2015 Jun 9. PMID 26060122
- [Derived] Montalescot G, Collet JP, Ecollan P, Bolognese L, Ten Berg J, Dudek D, Hamm C, Widimsky P, Tanguay JF, Goldstein P, Brown E, Miller DL, LeNarz L, Vicaut E; ACCOAST Investigators. Effect of prasugrel pre-treatment strategy in patients undergoing percutaneous coronary intervention for NSTEMI: the ACCOAST-PCI study. J Am Coll Cardiol. 2014 Dec 23;64(24):2563-2571. doi: 10.1016/j.jacc.2014.08.053. PMID 25524333
- [Derived] Montalescot G, Bolognese L, Dudek D, Goldstein P, Hamm C, Tanguay JF, ten Berg JM, Miller DL, Costigan TM, Goedicke J, Silvain J, Angioli P, Legutko J, Niethammer M, Motovska Z, Jakubowski JA, Cayla G, Visconti LO, Vicaut E, Widimsky P; ACCOAST Investigators. Pretreatment with prasugrel in non-ST-segment elevation acute coronary syndromes. N Engl J Med. 2013 Sep 12;369(11):999-1010. doi: 10.1056/NEJMoa1308075. Epub 2013 Sep 1. PMID 23991622
- [Derived] Montalescot G, Bolognese L, Dudek D, Goldstein P, Hamm C, Tanguay JF, ten Berg J, Widimsky P, Luo J, Miller DL, Goedicke J. A comparison of prasugrel at the time of percutaneous coronary intervention or as pretreatment at the time of diagnosis in patients with non-ST-segment elevation myocardial infarction: design and rationale for the ACCOAST study. Am Heart J. 2011 Apr;161(4):650-656.e1. doi: 10.1016/j.ahj.2010.10.017. Epub 2011 Feb 25. PMID 21473962

RESULTS

PARTICIPANT FLOW:
Groups:
- Non Pre-treatment: A placebo oral loading dose (LD) was given at the time of diagnosis and a 60 milligrams (mg) oral LD of prasugrel was given at the time of percutaneous coronary intervention (PCI) followed by 5 mg or 10 mg oral daily maintenance dose of prasugrel for 30 days.
- Pre-treatment: A 30 mg oral LD of prasugrel was given at diagnosis and a 30 mg oral dose of prasugrel was given at the time of PCI followed by 5 mg or 10 mg oral daily maintenance dose of prasugrel for 30 days.
Period: Overall Study
Arm/Group | Non Pre-treatment | Pre-treatment
Started | 1996 | 2037
Received at Least 1 Dose of Study Drug | 1996 | 2037
Completed | 1924 | 1958
Not Completed | 72 | 79
Not completed — Death | 21 | 16
Not completed — Adverse Event | 1 | 0
Not completed — Sponsor Decision | 3 | 7
Not completed — Physician Decision | 19 | 21
Not completed — Withdrawal by Subject | 14 | 19
Not completed — Entry Criteria not Met | 11 | 14
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non Pre-treatment | Pre-treatment | Total
Number analyzed (Participants) | 1996 | 2037 | 4033
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.59 (11.239) | 63.80 (11.270) | 63.69 (11.254)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 558 | 552 | 1110
  Male | 1438 | 1485 | 2923

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Occurrence of Cardiovascular (CV) Death, Myocardial Infarction (MI), Stroke, Urgent Revascularization (UR), or Glycoprotein (GP) IIb/IIIa Inhibitor Bailout
Description: The percentage of participants is the total number of participants experiencing a CV death, MI, stroke, UR or GPIIb/IIIa Inhibitor bailout divided by number of participants in the treatment arm multiplied by 100. Endpoint events were adjudicated by the Clinical Endpoint Committee.
Time Frame: First loading dose (LD) through 7 days after first LD
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Non Pre-treatment: A placebo oral LD was given at the time of diagnosis and a 60 milligrams (mg) oral LD of prasugrel was given at the time of percutaneous coronary intervention (PCI) followed by 5 mg or 10 mg oral daily maintenance dose of prasugrel for 30 days.
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 1996 | 2037
percentage of participants | 9.77 | 9.97

2. Secondary Outcome: Percentage of Participants With All-Cause Death, Myocardial Infarction (MI), Stroke, or All Coronary Artery Bypass Graft (CABG) and Non-CABG Thrombolysis in Myocardial Infarction (TIMI) Major Bleeding
Description: The percentage of participants is the total number of participants experiencing an all-cause death, MI, stroke or CABG and non-CABG TIMI major bleeding divided by number of participants in the treatment arm multiplied by 100. Endpoint events were adjudicated by the Clinical Endpoint Committee.
Time Frame: First loading dose (LD) through 7 days after first LD
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Non Pre-treatment: A placebo LD was given at the time of diagnosis and a 60 milligrams (mg) oral LD of prasugrel was given at the time of percutaneous coronary intervention (PCI) followed by 5 mg or 10 mg oral daily maintenance dose of prasugrel for 30 days.
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 1996 | 2037
percentage of participants | 7.57 | 8.64

3. Secondary Outcome: Percentage of Participants With Incidence of Cardiovascular (CV) Death, Myocardial Infarction (MI), or Stroke Through 30 Days From First Loading Dose (LD)
Description: The percentage of participants is the total number of participants experiencing a CV death, MI, or stroke divided by number of participants in the treatment arm multiplied by 100. Endpoint events were adjudicated by the Clinical Endpoint Committee.
Time Frame: First LD through 30 days after first LD
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 1996 | 2037
percentage of participants | 7.21 | 7.07

4. Secondary Outcome: Percentage of Participants With Incidence of Cardiovascular (CV) Death or Myocardial Infarction (MI) Through 30 Days From First Loading Dose (LD)
Description: The percentage of participants is the total number of participants experiencing a CV death or MI divided by number of participants in the treatment arm multiplied by 100. Endpoint events were adjudicated by the Clinical Endpoint Committee.
Time Frame: First LD through 30 days after first LD
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 1996 | 2037
percentage of participants | 6.51 | 6.63

5. Secondary Outcome: Percentage of Participants With Incidence of Cardiovascular (CV) Death, Myocardial Infarction (MI), or Urgent Revascularization (UR) Through 30 Days From First Loading Dose (LD)
Description: The percentage of participants is the total number of participants experiencing a CV death, MI, or UR divided by number of participants in the treatment arm multiplied by 100. Endpoint events were adjudicated by the Clinical Endpoint Committee.
Time Frame: First LD through 30 days after first LD
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 1996 | 2037
percentage of participants | 7.31 | 7.71

6. Secondary Outcome: Percentage of Participants With Incidence of Cardiovascular (CV) Death Through 30 Days From First Loading Dose (LD)
Description: The percentage of participants is the total number of participants experiencing a CV death divided by number of participants in the treatment arm multiplied by 100. Endpoint events were adjudicated by the Clinical Endpoint Committee.
Time Frame: First LD through 30 days after first LD
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 1996 | 2037
percentage of participants | 1.10 | 0.69

7. Secondary Outcome: Percentage of Participants With Incidence of Definite or Probable Stent Thrombosis (ST) According to the Academic Research Consortium (ARC) Criteria Through 30 Days From First Loading Dose (LD)
Description: ARC criteria were used to define ST. Definite ST is angiographic or pathologic confirmation of partial or total thrombotic occlusion within the peri-stent region, and at least one of the following additional criteria: acute ischemic symptoms; ischemic electrocardiogram changes; elevated cardiac biomarkers. Probable ST is any unexplained death within 30 days of stent implantation; any MI, which is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of ST and in the absence of any other obvious cause. The percentage of participants is the total number of participants experiencing a definite or probable stent thrombosis divided by number of participants in the treatment arm multiplied by 100. Endpoint events were adjudicated by the Clinical Endpoint Committee.
Time Frame: First LD through 30 days after first LD
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 1996 | 2037
percentage of participants | 0.25 | 0.10

8. Secondary Outcome: Percentage of Participants With All-cause Death, Myocardial Infarction (MI), Stroke, or All Coronary Artery Bypass Graft (CABG) and Non-CABG Thrombolysis in Myocardial Infarction (TIMI) Major Bleeding Through 30 Days From First Loading Dose (LD)
Description: as for outcome 2
Time Frame: First LD through 30 days after first LD
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 1996 | 2037
percentage of participants | 8.52 | 9.47

9. Secondary Outcome: Change in Standardized Troponin From Baseline to Percutaneous Coronary Intervention (PCI)
Description: Standardized troponin is defined as the ratio of the assayed troponin value divided by the upper limit of normal (ULN). Least Squares (LS) means were obtained from an Analysis of Covariance (ANCOVA) model with treatment as a fixed effect and baseline standardized troponin as a covariate.
Time Frame: Baseline, before PCI (not greater than 48 hours after randomization)
Population: All randomized participants who received at least 1 dose of study drug, had standardized troponin measured at baseline and before PCI (not greater than 48 hours after randomization).
Measure: Least Squares Mean (Standard Error); unit: ratio of assayed troponin/ULN
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 454 | 511
ratio of assayed troponin/ULN | -11.24 (8.93) | 2.82 (8.42)

10. Secondary Outcome: Percentage of Participants With Incidence of All Coronary Artery Bypass Graft (CABG) or Non-CABG Thrombolysis In Myocardial Infarction (TIMI) Major Bleeding
Description: The percentage of participants is the total number of participants experiencing a CABG or non-CABG TIMI major bleeding divided by number of participants in the treatment arm multiplied by 100. Endpoint events were adjudicated by the Clinical Endpoint Committee.
Time Frame: First loading dose (LD) through 7 days after first LD
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 1996 | 2037
percentage of participants | 1.35 | 2.55

11. Other Pre Specified Outcome: Summary of All-Cause Death
Description: All deaths, regardless of possible relatedness, were adjudicated by the Clinical Endpoint Committee (CEC) and are reported in this table.
Time Frame: Randomization through 30 days
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Non Pre-treatment | Pre-treatment
Number analyzed (Participants) | 1996 | 2037
participants
  Congestive Heart Failure | 1 | 0
  Cardiogenic Shock | 5 | 5
  During or Immediately Following a CABG Procedure | 5 | 1
  During or Immediately Following a PCI Procedure | 2 | 1
  Myocardial Infarction | 2 | 1
  Dysrhythmia | 0 | 1
  Sudden Cardiac Death | 4 | 1
  Intracranial Hemorrhage | 1 | 1
  Stroke, non-hemorrhagic | 0 | 1
  Other Cardiovascular | 2 | 2
  Non-Cardiac Hemorrhage, Not Intracranial | 0 | 1
  Infection | 1 | 0
  Cancer | 0 | 1

ADVERSE EVENTS:
Arm/Group | Non Pre-treatment | Pre-treatment
Serious Adverse Events (participants affected / at risk) | 167/1996 | 206/2037
Other Adverse Events (participants affected / at risk) | 860/1996 | 876/2037
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non Pre-treatment (N=1996) | Pre-treatment (N=2037)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperchromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 6 (6)
Angina pectoris (Cardiac disorders) | 1 (1) | 5 (6)
Angina unstable (Cardiac disorders) | 2 (2) | 6 (6)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 3 (3)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bifascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 3 (3) | 5 (5)
Cardiac failure (Cardiac disorders) | 4 (4) | 3 (4)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 5 (5) | 7 (7)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 2 (2) | 3 (3)
Coronary artery embolism (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery thrombosis (Cardiac disorders) | 4 (4) | 5 (5)
Coronary no-reflow phenomenon (Cardiac disorders) | 1 (1) | 0 (0)
Coronary ostial stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Haemorrhage coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 10 (10) | 15 (15)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial rupture (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 4 (4) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis constrictive (Cardiac disorders) | 1 (1) | 0 (0)
Pleuropericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Postinfarction angina (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 5 (5) | 7 (7)
Ventricular flutter (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 4 (4) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 5 (5)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 2 (2)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 8 (8) | 9 (9)
Device dislocation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
Puncture site haemorrhage (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Spinal pain (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Thrombosis in device (General disorders) | 4 (5) | 1 (1)
Vessel puncture site haematoma (General disorders) | 2 (2) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 2 (2)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4)
Puncture site infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Vena cava injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Cardiac output decreased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 2 (2)
Inflammatory marker increased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 2 (2)
Troponin t increased (Investigations) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 2 (2)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 2 (2)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 5 (5) | 6 (6)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 10 (10) | 16 (17)
Thrombolysis (Surgical and medical procedures) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arterial rupture (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 3 (3) | 6 (6)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Non Pre-treatment (N=1996) | Pre-treatment (N=2037)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 17 (17)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
Accelerated idioventricular rhythm (Cardiac disorders) | 3 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Angina pectoris (Cardiac disorders) | 18 (19) | 14 (15)
Angina unstable (Cardiac disorders) | 6 (6) | 4 (4)
Aortic valve incompetence (Cardiac disorders) | 5 (5) | 5 (5)
Aortic valve sclerosis (Cardiac disorders) | 0 (0) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 3 (3) | 3 (3)
Arrhythmia (Cardiac disorders) | 2 (2) | 3 (3)
Arrhythmia supraventricular (Cardiac disorders) | 3 (3) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 28 (28) | 36 (38)
Atrial flutter (Cardiac disorders) | 5 (5) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 2 (2) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 6 (6)
Bradycardia (Cardiac disorders) | 21 (21) | 25 (25)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 21 (21) | 15 (15)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 4 (4)
Coronary artery dissection (Cardiac disorders) | 3 (3) | 1 (1)
Coronary artery embolism (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 6 (6)
Coronary artery perforation (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 2 (2)
Coronary artery thrombosis (Cardiac disorders) | 3 (3) | 7 (7)
Coronary no-reflow phenomenon (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 6 (6)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 17 (17) | 19 (19)
Myocardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 49 (50) | 41 (41)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 3 (3) | 2 (2)
Palpitations (Cardiac disorders) | 7 (7) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)
Pericarditis (Cardiac disorders) | 3 (3) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 3 (3)
Tachyarrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 7 (7)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 10 (10) | 6 (6)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 4 (4) | 5 (5)
Ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 10 (12) | 16 (16)
Gene mutation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Right aortic arch (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Type v hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 3 (3)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 11 (11)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 4 (4)
Hypothyroidism (Endocrine disorders) | 4 (4) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 2 (2) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Eye oedema (Eye disorders) | 1 (1) | 0 (0)
Panophthalmitis (Eye disorders) | 1 (1) | 0 (0)
Refraction disorder (Eye disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 12 (12)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (11) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 19 (19) | 19 (19)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 6 (6)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gingival bleeding (Gastrointestinal disorders) | 9 (9) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 5 (5) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 3 (3)
Mesenteric haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 22 (22) | 25 (25)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 10 (10) | 9 (9)
Asthenia (General disorders) | 17 (17) | 15 (15)
Catheter site discharge (General disorders) | 0 (0) | 1 (1)
Catheter site erythema (General disorders) | 2 (2) | 0 (0)
Catheter site haematoma (General disorders) | 6 (6) | 5 (5)
Catheter site haemorrhage (General disorders) | 5 (5) | 7 (8)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 2 (2) | 0 (0)
Catheter site phlebitis (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 6 (6) | 6 (6)
Chest pain (General disorders) | 55 (56) | 47 (50)
Chills (General disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 1 (1)
Drug intolerance (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 3 (3) | 9 (9)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Hypertrophy (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 2 (2)
Injection site haemorrhage (General disorders) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Oedema (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 9 (9) | 14 (15)
Pain (General disorders) | 4 (4) | 2 (2)
Polyp (General disorders) | 0 (0) | 1 (1)
Puncture site discharge (General disorders) | 1 (1) | 0 (0)
Puncture site haemorrhage (General disorders) | 2 (2) | 7 (7)
Puncture site pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 24 (24) | 33 (33)
Spinal pain (General disorders) | 2 (2) | 3 (3)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Thrombosis in device (General disorders) | 3 (3) | 0 (0)
Vessel puncture site haematoma (General disorders) | 9 (9) | 12 (12)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 4 (6)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 3 (3)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to chemicals (Immune system disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Iodine allergy (Immune system disorders) | 4 (4) | 2 (2)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 3 (3)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 3 (3) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Eye abscess (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Groin infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis a (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis e (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Leprosy (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 3 (3)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Nosocomial infection (Infections and infestations) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 10 (10) | 10 (10)
Viral diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1/552 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 14 (14) | 15 (16)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dislocation of sternum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 9 (9)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 5 (5) | 7 (7)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Procedural hypotension (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Antibiotic resistant staphylococcus test positive (Investigations) | 1 (1) | 0 (0)
Aortic bruit (Investigations) | 1 (1) | 1 (1)
Arteriogram coronary (Investigations) | 1 (1) | 0 (0)
Blood bilirubin decreased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 7 (7) | 6 (6)
Blood creatine phosphokinase mb increased (Investigations) | 4 (4) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1)
Blood glucose increased (Investigations) | 2 (2) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 4 (4)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Blood urine (Investigations) | 1 (2) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 2 (2) | 2 (2)
C-reactive protein increased (Investigations) | 1 (1) | 3 (3)
Carbohydrate tolerance decreased (Investigations) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 16 (16) | 19 (19)
Cardiac murmur (Investigations) | 2 (2) | 3 (3)
Central venous pressure increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 2 (2) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0)
Electrocardiogram st segment depression (Investigations) | 1 (1) | 0 (0)
Electrocardiogram st segment elevation (Investigations) | 0 (0) | 1 (1)
Electrophoresis protein abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 20 (20) | 28 (28)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 5 (5)
Hepatitis c virus test positive (Investigations) | 1 (1) | 0 (0)
Inflammatory marker increased (Investigations) | 1 (1) | 1 (1)
Low density lipoprotein increased (Investigations) | 2 (2) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Peripheral pulse decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 2 (2)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1/1485 (1)
Transaminases increased (Investigations) | 1 (1) | 2 (2)
Troponin i increased (Investigations) | 4 (4) | 4 (4)
Troponin increased (Investigations) | 3 (3) | 4 (4)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 24 (24) | 27 (27)
Dyslipidaemia (Metabolism and nutrition disorders) | 27 (27) | 22 (22)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Gout (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 87 (87) | 72 (72)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 42 (42) | 26 (26)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Hypo hdl cholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (18) | 14 (14)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lipid metabolism disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Overweight (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 20 (20)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (14) | 17 (17)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Akinesia (Nervous system disorders) | 1 (2) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 3 (3) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 3 (3) | 4 (4)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 11 (11) | 14 (14)
Drop attacks (Nervous system disorders) | 1 (2) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 48 (48) | 44 (45)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 8 (8) | 10 (10)
Psychomotor hyperactivity (Nervous system disorders) | 2 (2) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 5 (5) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 3 (3)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 10 (10) | 13 (13)
Confusional state (Psychiatric disorders) | 0 (0) | 6 (6)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 4 (4) | 3 (3)
Disorientation (Psychiatric disorders) | 2 (2) | 3 (4)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Histrionic personality disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3)
Libido disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Transient psychosis (Psychiatric disorders) | 2 (2) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 4 (4)
Haematuria (Renal and urinary disorders) | 6 (6) | 9 (9)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal failure (Renal and urinary disorders) | 9 (9) | 8 (8)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure chronic (Renal and urinary disorders) | 6 (6) | 5 (5)
Strangury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (5) | 2 (2)
Balanoposthitis (Reproductive system and breast disorders) | 1/1438 (1) | 0/1485 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/1438 (0) | 2/1485 (2)
Breast haematoma (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 1/1438 (1) | 0/1485 (0)
Epididymitis (Reproductive system and breast disorders) | 1/1438 (1) | 0/1485 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 4/1438 (4) | 1/1485 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1/1438 (1) | 1/1485 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0/558 (0) | 2/552 (2)
Penis disorder (Reproductive system and breast disorders) | 0/1438 (0) | 1/1485 (1)
Prostatic calcification (Reproductive system and breast disorders) | 1/1438 (1) | 0/1485 (0)
Testicular oedema (Reproductive system and breast disorders) | 0/1438 (0) | 1/1485 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/558 (1) | 2/552 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 22 (22)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 21 (21)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 28 (30) | 38 (48)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 12 (12) | 10 (12)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 11 (11) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 13 (13) | 4 (4)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Xanthoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bladder catheter removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Blood product transfusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 3 (3)
Carotid angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 2 (2) | 5 (5)
Coronary revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Dialysis (Surgical and medical procedures) | 0 (0) | 1 (1)
Heart valve operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Packed red blood cell transfusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 14 (14) | 8 (8)
Platelet transfusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Thromboembolectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic calcification (Vascular disorders) | 1 (1) | 0 (0)
Aortic dilatation (Vascular disorders) | 1 (1) | 3 (3)
Aortic disorder (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 5 (5) | 3 (3)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 57 (62) | 96 (97)
Haemodynamic instability (Vascular disorders) | 2 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 10 (10) | 13 (13)
Hypertension (Vascular disorders) | 88 (88) | 90 (90)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 23 (23) | 28 (29)
Ischaemia (Vascular disorders) | 2 (2) | 1 (1)
Macroangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (4) | 4 (4)
Peripheral artery dissection (Vascular disorders) | 0 (0) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 2 (2)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 4 (4) | 3 (3)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 1 (1)
Reperfusion injury (Vascular disorders) | 3 (3) | 3 (3)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 6 (7) | 4 (4)
Varicose vein ruptured (Vascular disorders) | 0 (0) | 1 (1)
Vascular occlusion (Vascular disorders) | 2 (2) | 1 (1)
Vasospasm (Vascular disorders) | 2 (3) | 2 (2)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days